CLINICAL TRIAL: NCT03984396
Title: Optimal Medication Management in Alzheimer's Disease and Dementia
Acronym: Optimize
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Johns Hopkins University (Other); Duke University (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R33AG057289 (NIH)
Record Dates: First submitted 2019-05-24; First posted 2019-06-13 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Dementia
Keywords: dementia; cognitive impairment; multimorbidity/comorbidity; polypharmacy; deprescriptions; patient education; deprescribe
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A pragmatic cluster randomized educational intervention with a delayed control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Patient and Clinician (Experimental): Intervention educational materials provided to patient and family and clinician
  Interventions: Other: Educational Materials - Patient & Clinician
- Delayed Intervention (No Intervention): Usual care

INTERVENTIONS:
Other: Educational Materials - Patient & Clinician — deprescribing information for patient & clinician
  Arms: Intervention - Patient and Clinician

SUMMARY:
The study objective is to conduct a pragmatic deprescribing intervention for people with Alzheimer's Disease or Related Dementia with Multiple Chronic Conditions (ADRD-MCC) so that these patients are on 'just right' medication regimens.

The intervention will be a pragmatic, cluster randomized trial of medication optimization through increased awareness of deprescribing for the ADRD-MCC population. It will be delivered in primary care at the clinic level with a wait-list control design. As a pragmatic intervention it is designed to be relatively simple, have broad inclusion/exclusion criteria, and be implemented across the Kaiser Permanente Colorado (KPCO) system. The intervention will have two components: a patient/care partner component focused on education and activation about potential deprescribing including sending out a brochure, and a clinician component focused on increasing clinician awareness through monthly Tip Sheets about options and processes for deprescribing in the ADRD-MCC population linked to upcoming visits. The intervention will take place at 18 primary care offices in the Denver-Boulder service delivery area with 9 as initial intervention sites and 9 as delayed intervention sites.

DETAILED DESCRIPTION:
The study objective is to conduct a pragmatic deprescribing intervention for people with Alzheimer's Disease or Related Dementia with Multiple Chronic Conditions (ADRD-MCC) so that these patients are on 'just right' medication regimens.

There are two components to the intervention: Patient/ care partner education and clinician education. Patient/care partner educational materials about medication optimization will be mailed to eligible members who have upcoming appointments with primary care physicians (PCPs) within 2 weeks of scheduled visits. The initial intervention period will run for 12 months and the delayed intervention period will run for 12 months. Primary care clinicians at the intervention clinics who care for adults (Internal Medicine [IM] and Family Medicine [FM]) will receive education on medication optimization and options for deprescribing through an initial presentation at a monthly team meeting at the beginning of the intervention period, as well as periodic Tip Sheet updates on managing deprescribing in specific situations. Primary care clinicians will receive notification via staff message when materials have been sent to patients with an upcoming appointment.

The intervention has two aims:

Aim 1: In a cluster randomized pragmatic trial, test the effectiveness of a primary care based, clinic level deprescribing intervention on two primary outcomes: number of chronic medications and number of potentially inappropriate medications (PIMs) among older adults with ADRD-MCC.

Aim 2: Evaluate the effect of the intervention on secondary outcomes of adverse drug events (falls, bleeding episodes, hypoglycemic episodes), reductions in dosage for selected PIMs (benzodiazepines, opioids, anti-psychotics), hospital, emergency department and skilled nursing facility utilization, and activities of daily living.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age>=65
* Bonded to a primary care physician (PCP) in the Kaiser Permanente Colorado (KPCO) - Denver-Boulder service area
* Diagnosis of Alzheimer's Dementia or Related Dementia or Mild Cognitive Impairment (MCI) from ICD-9 or ICD-10 visit codes or from the problem list in the Electronic Health Record (EHR)
* One or more additional chronic conditions from a list of 86 chronic medical conditions
* Be taking 5 or more chronic medications (defined as a 28+ days' supply of medication on the eligibility date; excluding non-indicated medications such as vaccines and anesthetics based on 2-digit GPI codes
* Of this eligible population, those who have at least one visit with a PCP during the intervention period will receive the patient portion of the intervention.

Patient Exclusion Criteria:

* Individuals residing in long term care facilities or enrolled in hospice care at baseline
* Individuals residing at home but receiving all their primary care through the KPCO Complex Care Home Rounding service which replaces primary care delivery

Clinician Inclusion Criteria:

* PCP for adult patients in the KPCO Denver-Boulder service area.

Clinician Exclusion Criterion:

* PCP for adult patients at the Longmont Medical Office since Longmont was the pilot study site.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7398 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Number of chronic medications | 6 months post brochure mailing
  Number of chronic medications defined as those with at least a 28 days supply
Number of chronic medications | 12 months post brochure mailing
  Number of chronic medications defined as those with at least a 28 days supply
Number of potentially inappropriate medications | 6 months post brochure mailing
  Number of chronic medications that are listed as potentially inappropriate for older adults based on the Beers list.
Number of potentially inappropriate medications | 12 months post brochure mailing
  Number of chronic medications that are listed as potentially inappropriate for older adults based on the Beers list.

SECONDARY OUTCOMES:
Treatment change | 12 months post initial brochure mailing
  Change in dose from baseline to outcome measurement for selected medications: benzodiazepines, opioids, antipsychotics
Selected adverse drug event (ADE) rates | 12 months post brochure mailing
  Three types of ADEs: falls; hemorrhagic events; and episodes of hypoglycemia in individuals with diabetes.
Hospitalization Rate, Skilled Nursing Facility Admissions Rate, Emergency Department Visit Rate | 12 months post brochure mailing
  Presence/ absence of a one of these admissions over the year prior to baseline and post intervention. (We will distinguish between temporary and permanent admissions to skilled nursing facilities.)
Activities of daily living as reported in the Medicare Health Risk Assessment (MHRA) | 3 days to 365 days after a participant's study index date
  Activities of Daily Living are reported by patients/ proxy responders as part of the annual MHRA. These data will be available on the subset of participants who have completed the MHRA. Data from the most recent MHRA will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reeve E, Bayliss EA, Shetterly S, Maiyani M, Gleason KS, Norton JD, Sheehan OC, Green AR, Maciejewski ML, Drace M, Sawyer J, Boyd CM. Willingness of older people living with dementia and mild cognitive impairment and their caregivers to have medications deprescribed. Age Ageing. 2023 Jan 8;52(1):afac335. doi: 10.1093/ageing/afac335. PMID 36702513
- [Background] Bayliss EA, Shetterly SM, Drace ML, Norton JD, Maiyani M, Gleason KS, Sawyer JK, Weffald LA, Green AR, Reeve E, Maciejewski ML, Sheehan OC, Wolff JL, Kraus C, Boyd CM. Deprescribing Education vs Usual Care for Patients With Cognitive Impairment and Primary Care Clinicians: The OPTIMIZE Pragmatic Cluster Randomized Trial. JAMA Intern Med. 2022 May 1;182(5):534-542. doi: 10.1001/jamainternmed.2022.0502. PMID 35343999
- [Background] Green AR, Boyd CM, Gleason KS, Wright L, Kraus CR, Bedoy R, Sanchez B, Norton J, Sheehan OC, Wolff JL, Reeve E, Maciejewski ML, Weffald LA, Bayliss EA. Designing a Primary Care-Based Deprescribing Intervention for Patients with Dementia and Multiple Chronic Conditions: a Qualitative Study. J Gen Intern Med. 2020 Dec;35(12):3556-3563. doi: 10.1007/s11606-020-06063-y. Epub 2020 Jul 29. PMID 32728959
- [Background] Bayliss EA, Shetterly SM, Drace ML, Norton J, Green AR, Reeve E, Weffald LA, Wright L, Maciejewski ML, Sheehan OC, Wolff JL, Gleason KS, Kraus C, Maiyani M, Du Vall M, Boyd CM. The OPTIMIZE patient- and family-centered, primary care-based deprescribing intervention for older adults with dementia or mild cognitive impairment and multiple chronic conditions: study protocol for a pragmatic cluster randomized controlled trial. Trials. 2020 Jun 18;21(1):542. doi: 10.1186/s13063-020-04482-0. PMID 32552857
- [Background] Sheehan OC, Gleason KS, Bayliss EA, Green AR, Drace ML, Norton J, Reeve E, Shetterly SM, Weffald LA, Sawyer JK, Maciejewski ML, Kraus C, Maiyani M, Wolff J, Boyd CM. Intervention design in cognitively impaired populations-Lessons learned from the OPTIMIZE deprescribing pragmatic trial. J Am Geriatr Soc. 2023 Mar;71(3):774-784. doi: 10.1111/jgs.18148. Epub 2022 Dec 12. PMID 36508725
- [Background] Orla Sheehan and others, Intervention Design With Cognitively Impaired Populations: The Optimize Deprescribing Intervention, Innovation in Aging, Volume 5, Issue Supplement_1, 2021, Page 401, https://doi.org/10.1093/geroni/igab046.1558
- [Background] Green AR, Weffald LA, Powers JD, Drace ML, Norton JD, Boyd CM, Bayliss EA. Assessing medication appropriateness as a deprescribing outcome. J Am Geriatr Soc. 2023 Dec;71(12):3918-3920. doi: 10.1111/jgs.18562. Epub 2023 Aug 26. No abstract available. PMID 37632424
- [Background] Boyd CM, Shetterly SM, Powers JD, Weffald LA, Green AR, Sheehan OC, Reeve E, Drace ML, Norton JD, Maiyani M, Gleason KS, Sawyer JK, Maciejewski ML, Wolff JL, Kraus C, Bayliss EA. Evaluating the Safety of an Educational Deprescribing Intervention: Lessons from the Optimize Trial. Drugs Aging. 2024 Jan;41(1):45-54. doi: 10.1007/s40266-023-01080-y. Epub 2023 Nov 20. PMID 37982982